CLINICAL TRIAL: NCT04441047
Title: Safety and Efficacy of ALLOSTIM® Universal Anti-Viral Immunodulatory Vaccine for Healthy Elderly Adults
Brief Title: Universal Anti-Viral Vaccine for Healthy Elderly Adults
Acronym: ALLOPRIME
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mirror Biologics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MBI-001-ALLOPRIME
Record Dates: First submitted 2020-06-17; First posted 2020-06-22 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Virus Diseases; Pneumonia; COVID-19 Respiratory Infection; RSV Pneumonia; Influenza, Human; ARDS, Human
Keywords: universal viral vaccine; COVID-19; AlloStim; elderly
MeSH Terms: conditions — Virus Diseases; Pneumonia; Influenza, Human; Respiratory Distress Syndrome; COVID-19

STUDY DESIGN:
Intervention Model Description: Subjects over 65yo in two cohorts: ages 65-74 and age 75+
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Vaccination (Experimental): ID injection AlloStim Days 0, 3/4, 7, 10/11 and 14
  Interventions: Drug: AlloStim

INTERVENTIONS:
Drug: AlloStim — Living, activated allogeneic Th1-like memory immune cells

SUMMARY:
This protocol tests the safety and efficacy of a novel universal vaccine concept called "allo-priming" which is designed to protect elderly adults from progression of any type of viral infection, including possible protection against progression of the current outbreak of COVID-19 infection, and any future variants, strains, mutations of the causative SARS-CoV-2 virus as well as protection from any future currently unknown newly emergent novel viruses.

DETAILED DESCRIPTION:
The proposed Allo-Prime universal viral protection mechanism involves vaccination with a bioengineered living allogeneic cellular vaccine (AlloStim) derived from healthy blood donors. The vaccine is designed to create high titers of memory immune cells that are specific to the foreign antigens in the living cell vaccine. Upon encounter with any type of virus, these memory immune cells are activated and release cytokines including an immediate release of IFN-ϒ. This non-specific activation causes immune conditions similar to the conditions that occur in healthy younger patients that leads to rapid viral clearance and viral-specific memory immune response to clear infection and protect against recurrence.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females who are at least 65 years of age at time of enrollment
2. Good general health *
3. Clinical screening laboratory evaluations (white blood cell (WBC), hemoglobin (Hgb), platelets (PLTs), alanine transaminase (ALT), aspartate transaminase (AST), creatinine (Cr), alkaline phosphatase (ALP), total bilirubin (T. Bili), prothrombin time (PT), and partial thromboplastin time (PTT)) are within acceptable normal reference ranges at the clinical laboratory being used.
4. Normal EKG
5. Available for the duration of the study
6. Peripheral veins suitable for blood draw
7. Able to provide consent

Exclusion Criteria:

* 1. History of autoimmune disease 2. Currently being treated for cancer (other than non-melanoma skin cancer) 3. History of COPD 4. Any clinical condition requiring systemic steroids or any current immunosuppressive therapy 5. HIV positive or any other type of immunodeficiency disorder 6. History of cardiac disease: congestive heart failure > NYHA class 2; cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or Digoxin are permitted) 7. Uncontrolled hypertension defined as SBP ≥130 and/or DBP ≥ 80 mm Hg 8. Active clinically serious infections (> grade 2 CTCAE) 9. History of organ transplant or tissue allograft 10. Oral temperature ≥99.0 degrees Fahrenheit (37.2 degrees Celsius). 11. Pulse < 60 or >100 beats per minute. 12. Oxygen saturation <96% 13. Uncontrolled concurrent serious medical or psychiatric illness 14. History of blood transfusion reactions 15. Receipt of any type of influenza vaccine or COVID19 vaccine last dose within two weeks of planned first study drug injection (influenza vaccination after day 28 is permitted)

  * As determined by medical history and physical examination to evaluate acute or ongoing chronic medical diagnoses/conditions that have been present for at least 90 days, which would affect the assessment of safety of subjects. Chronic medical diagnoses/conditions should be stable for the last 60 days (no hospitalizations, emergency room (ER), or urgent care for condition or need for supplemental oxygen). This includes no change in chronic prescription medication, dose, or frequency as a result of deterioration of the chronic medical diagnosis/condition in the 60 days before enrollment. Any prescription change that is due to change of health care provider, insurance company, etc., or done for financial reasons, and in the same class of medication, will not be considered a deviation of this inclusion criterion. Any change in prescription medication due to improvement of a disease outcome, as determined by the participating site principal investigator (PI) or appropriate sub-investigator, will not be considered a deviation of this inclusion criterion.

Subjects may be on chronic or as needed (prn) medications if, in the opinion of the participating site PI or appropriate sub-investigator, they pose no additional risk to subject safety or assessment of reactogenicity and immunogenicity, and do not indicate a worsening of medical diagnosis/condition. Similarly, medication changes subsequent to enrollment and study vaccination are acceptable provided the change was not precipitated by deterioration in the chronic medical condition, and there is no anticipated additional risk to the subject or interference with the evaluation of responses to study vaccination.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
frequency of vaccine events | day 0 to day 28
  vaccine events such as fever, rash, abnormal vital signs
Proportion of subjects with positive T-cell response | day 0 to 1 year
  measurement of Th1/Th2 balance, allo-specific Th1/CTL response
Proportion of subjects able to suppress viral propagation | day 0 to 1 year
  ex-vivo challenge of blood samples with live virus including SARS-CoV-2, influenza A and B

CONTACTS AND LOCATIONS:
Overall Officials: Michael Har-Noy, MD, Study Director — Mirror Biologics, Inc.
Locations (4):
- United States (4):
  - Delray Physician Care Center, Delray Beach, Florida
  - Coral Research Clinic & Coral Diagnostic, Miami, Florida
  - Model Research, Tampa, Florida
  - Florida Medical Clinic, LLC, Zephyrhills, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Har-Noy M, Or R. Allo-priming as a universal anti-viral vaccine: protecting elderly from current COVID-19 and any future unknown viral outbreak. J Transl Med. 2020 May 12;18(1):196. doi: 10.1186/s12967-020-02363-3. PMID 32398026
- [Derived] Liu C, Yang X, Paoli-Bruno J, Sikes D, Marin-Ruiz AV, Thomas N, Shane R, Har-Noy M. Allo-Priming Reverses Immunosenescence and May Restore Broad Respiratory Viral Protection and Vaccine Responsiveness to the Elderly: Results of a Phase I/II Clinical Trial. Vaccines (Basel). 2025 Apr 25;13(5):463. doi: 10.3390/vaccines13050463. PMID 40432075
- See also: sponsor website — http://www.mirrorbio.com